CLINICAL TRIAL: NCT02023138
Title: Evaluation of the Acceptability, Feasibility and Effectiveness of Two Methods of Involvement of Patients With Cognitive Disability in Clinical Guidelines Development: a Randomized Crossover Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marie-Eve Lamontagne, Assistant professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: KT Canada 87776
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Brain Injury
Keywords: Clinical practice guideline; Brain injury; Acceptability; Feasibility; Effectiveness
MeSH Terms: conditions — Brain Injuries | interventions — Focus Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Focus group (Active Comparator)
  Interventions: Other: Focus group; Other: Wiki
- Wiki (Experimental)
  Interventions: Other: Focus group; Other: Wiki

INTERVENTIONS:
Other: Focus group — Two hours focus group to allow the participants to modify a clinical practice guideline recommendation
Other: Wiki — A specially tailored interactive communication website (Wiki) to allow the participants to modify a clinical practice guideline recommendation

SUMMARY:
There is a lack of evidence about the best method to involve the patient and population (IPP) into clinical practice guidelines (CPG) development. The goal of this pilot study is to document the acceptability, feasibility and effectiveness of two methods for the implication of patients with a traumatic brain injury (TBI) in CPG development. Method: A single blind, randomized crossover trial will be performed with patients having a TBI. Participants: A convenience sample of 20 patients a) with a moderate-to-severe TBI (Glascow Coma Scale <13), b) living with a TBI for two to four years, c) French-speaking, d) able to use a computer and e) able to participate in a two-hour group meeting will be recruited among the members of the Associations TCC Des Deux Rives. Procedures: The patients will first receive a in-person training on guidelines and IPP. They will be randomized into Group 1 or Group 2 by a researcher blinded to experimentation. They will experiment either group discussion (control intervention) or a Wiki (experimental intervention). Phase 1: A week after the training, Group 1 participants will be invited to a discussion group animated by an experimented moderator, where they will be asked to discuss a CPG recommendation chosen by the research team in an existing CPG. The participants will be asked : 1) about their opinion of the recommendation; 2) if they have a preference in regard to the recommendation ; 3) if they have some modification, correction or addition to bring to this recommendation. In the mean time, Group 2 participants will receive an email presenting a link to a Wiki. They will be invited to answer the same three questions as Group 1, but using a Wiki platform. The patients will have a week to interact and answer the questions; recalls could be sent by email if required. At the end of Phase 1, participants of both groups will fill a questionnaire documenting the acceptability of the method experimented. Phase 2: As per the crossover design, the Group 1 participants will then be assigned to the Wiki intervention and the Group 2 participants will be assigned to the discussion group intervention. The procedure will be repeated with a second recommendation. At the end of Phase 2, the patients will be asked to answer a short survey to validate their preferences about the two methods. Tools: The acceptability of the methods will be evaluated with a questionnaire adapted from Sidani and al. and validated with three TBI individuals. The feasibility of the intervention will be evaluated using a) the number of participants who reached the group or the Wiki, b) the number of participants who completed the intervention c) the number of support interventions required in the group and in the Wiki. The effectiveness of the two methods will be evaluated by submitting the adapted recommendations to a panel of expert clinicians evaluators blinded to the methodologies of recommendations adaptation. They will be invited to rate the clarity, accuracy, appropriateness and usefulness of the recommendations. Analysis: Feasibility indicators will be reported using descriptive statistics. Within-subject analysis using non-parametric statistics will be performed to assess the acceptability of the two methods. AC1 coefficient of raters' agreement will be calculated on the expert evaluation scores, and the effectiveness of the methods will be compared using appropriate non parametric statistics to. Impact: This pilot trial will be the first one to evaluate methodologies for involving disabled individuals into CPG development.

ELIGIBILITY:
Inclusion Criteria:

* having suffered a moderate-to-severe TBI (Glascow Coma Scale <13)
* living with a TBI for two to four years
* French-speaking
* able to use a computer
* able to participate in a two-hour group meeting

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Immediatly (less than 12 hours) after the intervention, at the end of week 2 and week 3.
  The acceptability of the method will be evaluated through individual questionnaire administred seven days after having make the wiki available, or immediatly after the focus group.
Feasibility | At the end of the experimentation of the two methods (end of week 3)
  The feasability will be assed by considering the number of participants reaching and using each method, and by recording the number of support intervention required for the use of each method.
Effectiveness | Within one month after the experimentation of the two methods.
  After the adaptation of the two recommendations using the two methods, twenty experts, blind to the method used to formulate the recommendations, will rate each recommendation for its clarity, accuracy, appropriateness and usefulness of the recommendations using 10 points likert scales. An electronic questionnaire will be send to the experts and they will have one week to rate the recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Association de personnes TCC du Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Lamontagne ME, Gagnon MP, Perreault K, Gauthier V. Evaluating the Acceptability, Feasibility, and Outcomes of Two Methods Involving Patients With Disability in Developing Clinical Guidelines: Crossover Pilot Study. J Particip Med. 2021 Nov 23;13(3):e24319. doi: 10.2196/24319. PMID 34812733